CLINICAL TRIAL: NCT01419028
Title: A Retrospective, Non-interventional Epidemiologic Study of the Natural History of Patients With Severe Perinatal and Infantile Hypophosphatasia (HPP)
Brief Title: A Retrospective Study of the Natural History of Patients With Severe Perinatal and Infantile Hypophosphatasia (HPP)
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ENB-011-10
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia (HPP)
Keywords: Hypophosphatasia; HPP; Bone disease; Soft bones; Low alkaline phosphatase; Genetic metabolic disorder; Alkaline phosphatase; Tissue non-specific alkaline phosphatase; Rickets; Osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with perinatal and/or infantile onset HPP: Patients with a confirmed diagnosis of perinatal or infantile onset hypophosphatasia (HPP)

SUMMARY:
This study aims to characterize the natural history of patients with severe perinatal or infantile onset HPP.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are no approved disease-modifying treatments for patients with this disease. There is also limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or legal guardian(s) must provide written informed consent prior to data abstraction, unless all of the following apply:
* The patient is deceased; AND
* The responsible IRB/IEC/REB does not require informed consent per a review of their documented local policies for collecting retrospective data on patients who are deceased; AND
* Written confirmation is received from the responsible IRB/IEC/REB confirming that the abstracted data can be analyzed and used to support regulatory filings by the Sponsor
* Patient must have a documented diagnosis of HPP as indicated by 1 or more of the following:
* Documented ALPL gene mutation(s)
* Serum alkaline phosphatase (ALP) below the age-adjusted normal range and either plasma pyridoxal 5'-phosphate (PLP) or urinary phosphoethanolamine (PEA) above the upper limit of normal
* Serum ALP below the age-adjusted normal range and HPP-related radiographic abnormalities on X-ray
* Patient must have onset of signs of HPP prior to 6 months of age and have documentation of 1 or more of the following characteristics of perinatal and infantile HPP:
* Respiratory compromise (up to and including respiratory failure) requiring institution of respiratory support measure(s), requiring medication(s) for management of symptom(s), and/or associated with other respiratory complications (e.g., pneumonia(s), respiratory tract infection(s))
* Pyridoxine (vitamin B6)-responsive seizures
* Rachitic chest deformity

Exclusion Criteria:

Patients will be excluded from study participation if they have 1 or more of the following exclusion criteria:

* Patient received treatment with asfotase alfa at any time prior to data abstraction
* Patient has clinically significant other disease

Both living and deceased patients will be considered for study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with perinatal and/or infantile onset HPP. Thirty-six patients were invasively ventilated or died, and 12 patients were censored.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University school of medicine, Indianapolis, Indiana
  - Shriners Hospital for Children, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Cook Children's Health Care System, Fort Worth, Texas
- Royal Children's Hospital, Parkville, Australia
- University of Manitoba Health Sciences Centre, Winnipeg, Canada
- Germany (2):
  - Universitatsmedizin Mainz, Villa, Mainz
  - Universitätsklinikum Würzburg Kinderklinik, Pädiatrische Infektiologie und Immunologie, Würzburg
- Hospital Infantil Universitario Nino Jesus Universidad autonoma de Madrid, Madrid, Spain
- National Taiwan University Hospital, Taipei, Taiwan
- Birmingham Childrens Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Whyte MP, Rockman-Greenberg C, Ozono K, Riese R, Moseley S, Melian A, Thompson DD, Bishop N, Hofmann C. Asfotase Alfa Treatment Improves Survival for Perinatal and Infantile Hypophosphatasia. J Clin Endocrinol Metab. 2016 Jan;101(1):334-42. doi: 10.1210/jc.2015-3462. Epub 2015 Nov 3. PMID 26529632
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between Sept 2012 and Apr 2013. 65 patients were screened and 48 were enrolled at 12 sites in 7 countries. Patients were recruited from investigational sites established at academic research and medical centers known to diagnose and/or treat patients with HPP. Both living and deceased patients were considered to partricipate.
Groups:
- Retrospective Observational: Patients with severe perinatal and/or infantile onset HPP (ie, where signs of the disease are present before 6 months of age).
Period: Overall Study
Arm/Group | Retrospective Observational
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Thirteen participants were alive at the time of data abstraction and were censored in the analysis
Arm/Group | Retrospective Observational
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age is only for subjects who are alive at the time of data abstraction
  weeks | 506.9 (319.24)
Age, Customized [Number; unit: weeks] — Age is only for subjects who are alive at the time of data abstraction
  weeks
    <=18 years | 10
    Between 18 and 65 years | 3
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Australia | 2
  Canada | 11
  Germany | 6
  Spain | 1
  Switzerland | 1
  Taiwan | 1
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Overall survival is defined as the time from birth to time of death.
Time Frame: Retrospective data collected on or before the data of abstraction.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Retrospective Observational
Number analyzed (Participants) | 48
days | 270.5 [155.0 to 428.0]

2. Secondary Outcome: Invasive Ventilator-free Survival Time
Description: Invasive ventilator-free survival is defined as the time during which the patient is alive and not invasively ventilated. For the purpose of this study, invasive ventilation is defined as mechanical ventilation via intubation of trachaeostomy.
Time Frame: Retrospective data collected on or before the date of abstraction.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Retrospective Observational
Number analyzed (Participants) | 48
days | 236 [78 to 300]

ADVERSE EVENTS:
Arm/Group | Retrospective Observational
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was an observational study and, as such, serious and/or other [non-serious] adverse events were not collected/assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in a multicenter study involves a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis. Therefore, PIs are subject to certain disclosure and publication limitations.